CLINICAL TRIAL: NCT03651037
Title: Physical Activity Platform to Improve Bone Health in Cancer Survivors
Acronym: THRIVORS+BH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thrivors Inc (Industry)
Collaborators: Oregon Health and Science University (Other); Masonic Cancer Center, University of Minnesota (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Cathy Skinner, Principal Investigator, Thrivors Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: THRIVORSBH-01; R43CA224412 (NIH)
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Breast Cancer; Physical Activity; Bone Health
Keywords: cancer; bone health; physical activity; technology platfrom
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thrivors+BH (Experimental): For Thrivors+BH, a module will be developed for users to input pain and energy levels, enabling real-time customization of exercise regimens. Modules of clinically validated bone health exercises with instructional videos will be developed. Additionally, users will be able upload and send videos of themselves exercising for feedback and assessment. This version will contain bone health educational content, mindfulness and nutrition resources.
  Interventions: Behavioral: Thrivors+BH
- Thrivors Basic (Experimental): A Thrivors Basic version that lacks customization and video content will be developed. This version will contain bone health educational content, mindfulness and nutrition resources.
  Interventions: Behavioral: Thrivors+BH

INTERVENTIONS:
Behavioral: Thrivors+BH — Digital health platform for breast cancer patients that measures adherence and engagement.
  Other Names: Thrivors

SUMMARY:
Cancer treatment-induced bone loss and the subsequent risk of fractures in both men and women impacts not just survivors' quality of life, but is also a significant burden on national health care. Clinical studies have reported that moderate-intensity resistance exercises prevent a decline in bone health in female cancer survivors, and that strength training may reduce complications associated with cancer such as fatigue, muscle wasting, and bone loss. Unfortunately, only a small percentage of women who have had cancer, engage in and adhere to a strength training exercise routine.

The investigators have developed an internet-based application, Thrivors, that guides cancer survivors through exercise routines with light-to-moderate strength training in the home setting, and connects them to survivorship resources. In this Phase I proposal, the investigators will develop and deploy an enhanced version, Thrivors+BH, that disseminates resistance training exercises specifically impacting bone health (BH), integrated with video-based interactive feedback and tracking of adherence to exercise routines.

The goal is to validate Thrivors+BH as a novel tool to bridge the gaps between cancer survivorship, physical activity, value-based care and health care organizations (providers and payers), to positively impact bone health in breast cancer survivors.

DETAILED DESCRIPTION:
Significance: Cancer treatment-induced bone loss and the subsequent risk of fractures in both men and women is a significant burden on national health care. The number of cancer survivors in the United States will reach 18 million by 2022 and by 2025, the projected burden of osteoporosis is $25.3 billion. Cancer patients treated with medications that lower hormone levels face an increased risk of fractures. Clinical studies report that moderate- intensity resistance exercises prevent a decline in bone health in female cancer survivors, and that strength training may reduce complications associated with cancer such as fatigue, muscle wasting, and bone loss. Unfortunately, only a small percentage of female cancer survivors engage in and adhere to a strength training exercise routine. Several factors account for this low level of engagement such as poor awareness of the benefits of exercise, lack of motivation, and the lack of affordable and easily accessible exercise programs designed for cancer survivors. Internet-based self-managed programs of exercises and guidance can potentially address these problems, and can be scaled for broader dissemination.

Innovation: The Thrivors internet-based platform seeks to shift the current paradigm of poor adherence to exercise by providing an affordable and accessible means of improving outcomes for cancer survivors. The proposed product, Thrivors+BH, will be a first-of-its-kind offering of clinically validated bone health exercises that can be customized to a cancer survivor's pain and energy levels, with several novel interactive feedback features. The product will also have supportive modules for connecting with a community of other users, mindfulness training, nutritional advice and a repository of educational information. The Thrivors platform is scalable, device-agnostic, and allows analysis of de-identified usage data. With commercialization potential for healthcare providers and health insurance payers, Thrivors provides a value-based care delivery model focused on outcomes. There are multiple important physiologic and psychosocial secondary conditions that could be positively impacted by the Thrivors platform. For this specific application, the investigators will focus on adherence to bone health exercises.

Hypothesis: The investigators hypothesized that breast cancer survivors' adherence to an exercise regimen for bone health can be improved by enhancing the interactive and customizable features of a cloud-based, device-agnostic delivery method. To test the hypothesis and to establish the technical feasibility of the product, the investigators propose the following specific aims:

Specific Aim 1: Develop an enhanced participant experience platform for bone health-specific exercises.

For Thrivors+BH, a module will be developed for participants to input pain and energy levels, enabling real-time customization of exercise regimens. Modules of clinically validated bone health exercises with instructional videos will be developed. Additionally, participants will be able upload and send videos of themselves exercising for feedback and assessment. A Thrivors Basic version that lacks customization and video content will be developed. Both versions will contain bone health educational content, mindfulness and nutrition resources. Milestones: Over a 2-month period, development, usability testing (assessing content, features, input controls, navigational ease and click-through capabilities) and refinement will be completed, to enable deployment in a randomized clinical trial.

Specific Aim 2: Measure participant adherence and engagement. The two versions of the platform will be deployed in a 20-week, two-arm randomized controlled trial of 50 breast cancer survivors. Adherence to exercise sessions (primary outcome) and platform usage will be measured by platform software, while user engagement (secondary outcomes) will be assessed by surveys. Milestones: Differences between primary and secondary outcomes for the control and intervention groups will be evaluated. Usage statistics, motivational responses and user feedback will be used to further refine platform features and content.

The outcomes of this study will help validate the utility of the Thrivors platform in improving cancer survivors' adherence and engagement to exercise routines that positively impact post-treatment recovery. In the near-term, the findings will inform the design of a 12-month Phase II study to evaluate changes in biomarkers of bone health. In the longer term, the project aligns with the business goal to disseminate the Thrivors platform to a larger population of male and female cancer survivors across ethnic/racial minority groups, rural populations, and low socioeconomic status groups. The project also aligns with the mission of the NCI to develop innovative technology and service delivery models that increase the adoption, uptake, and sustainability of evidence-based interventions to improve public health.

ELIGIBILITY:
Inclusion Criteria:

* Female participants diagnosed at 40 - 70 years with non-metastatic breast cancer.
* Able to provide written informed consent.
* Completed chemotherapy, undergoing adjuvant hormonal therapy.
* Not currently on a prescribed exercise plan and cleared for exercise by physician.
* Access to a smart phone (with a data plan), tablet, or computer (with internet access).
* Able and willing to comply with the protocol, including completion of all surveys.

Exclusion Criteria:

* Less than 4 weeks post-surgery.
* Diagnosis of osteoporosis.
* Currently participating in two or more 30-min. sessions/week of resistance or impact exercises.
* Specific condition(s) or diagnosis, both physical or psychological, or physical exam finding that precludes participation in a physical exercise program.
* Participant has hemodynamically significant heart disease (e.g., heart failure) or an arrhythmic heart condition requiring medical therapy.
* Employees or family members of the investigator, study site, or sponsor directly involved with study management.
* Participants who, in the opinion of the primary investigator, should not participate in the study.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Number of participants to complete exercise sessions and surveys | 20 weeks
  Changes in baseline from exercise naive to exercise activated as well as improvements in well-being survey, patient activation measures, and bone health awareness

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Skinner, MA, Principal Investigator — Thrivors Inc
Locations (1):
- Thrivors Inc, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No